CLINICAL TRIAL: NCT01298635
Title: Comparison of Combined Phacotrabeculectomy and Trabeculectomy Only in the Treatment of Primary Angle-closure Glaucoma
Brief Title: Comparison of Phacotrabeculectomy and Trabeculectomy in the Treatment of Primary Angle-closure Glaucoma (PACG)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: Ministry of Science and Technology (Ambiguous); Guangdong Province, Department of Science and Technology (Other Government)
Responsible Party: Jian Ge, Zhongshan Ophthalmic Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GJ-PACG-phacotrab/trab
Record Dates: First submitted 2011-02-17; First posted 2011-02-18 (Estimated); Last update posted 2011-02-18 (Estimated); Status verified 2004-11

CONDITIONS: Glaucoma, Angle-Closure; Cataract
Keywords: Primary angle-closure glaucoma; cataract; trabeculectomy; phacotrabeculectomy
MeSH Terms: conditions — Glaucoma, Angle-Closure; Cataract | interventions — Trabeculectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- trab (Active Comparator)
  Interventions: Procedure: trabeculectomy
- phacotrab (Active Comparator)
  Interventions: Procedure: combined phacotrabeculectomy

INTERVENTIONS:
Procedure: combined phacotrabeculectomy — trabeculectomy plus phacoemulsification with intraocular lens implantation
  Arms: phacotrab
Procedure: trabeculectomy
  Arms: trab

SUMMARY:
Primary angle closure glaucoma (PACG) is caused by contact between the iris and trabecular meshwork, which in turn obstructs outflow of the aqueous humor from the eye. This contact between iris and trabecular meshwork (TM) may gradually damage the function of the meshwork until it fails to keep pace with aqueous production, and the pressure rises, and at last the optic nerve is damaged, the vision may be lost in some severe cases. Therefore, ocular pressure reduction is the key to treat the disease and prevent blindness. Trabeculectomy is the most common conventional surgery performed for glaucoma. This allows fluid to flow out of the eye through this opening, resulting in lowered intraocular pressure(IOP) and the formation of a bleb or fluid bubble on the surface of the eye.

Cataract surgery is common in the elderly. Cataract surgery is the removal of the natural lens of the eye (also called "crystalline lens") that has developed an opacification, which is referred to as a cataract. Cataract extraction includes intracapsular cataract extraction, extra capsular cataract extraction & phacoemulsification, and phacoemulsification is the preferred method. It has been reported that IOP reduction could occur in cataract patients with PACG after the cataract surgery. For some cases with PACG, such IOP reduction may be insufficient for neuronal protection, and many patients still require glaucoma medication and incisional surgery such as trabeculectomy to control IOP. In such cases, a combined cataract-glaucoma procedure (phacotrabeculectomy) is a reasonable option. In keeping with this concept, previous studies have shown that phacotrabeculectomy could effectively and simultaneously reduce IOP and improve vision in patients with a coexistence of PACG and vision-threatening cataract. However, phacotrabeculectomy may heighten inflammatory response, result in a higher frequency of postoperative complications such as hyphema and fibrin in the anterior chamber, endophthalmitis, and increased scarring of the filtering bleb. Thus, it is unclear whether phacotrabeculectomy is as effective and safe as trabeculectomy in lowering IOP for PACG patients.

In the present study, the investigators compared the efficacy and safety of phacotrabeculectomy and trabeculectomy in patients with coexisting PACG and cataract.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of primary angle-closure glaucoma with co-existing cataract

Exclusion Criteria:

* secondary glaucoma
* history of any intraocular surgery, including laser iridectomy

Ages: 40 Years to 82 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2005-01; Primary Completion 2007-01 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
reduction of intraocular pressure | within 18 months after surgery
  the difference of intraocular pressure between preoperation and postopration at the last followup

SECONDARY OUTCOMES:
Number of Glaucoma medications | within 18 months after surgery
  to compare the number of pre- and post-operative intraocular pressure lowering drugs
Morphology of filtering blebs | within 18 months after surgery
  The filtering bleb morphology was assessed using simplified the Indiana bleb assessment grading system with a slit-lamp.Then to analyze the number of eyes with different type of blebs
Visual outcomes | within 18 months after surgery
  best corrected visual acuity was measured on Snellen decimal charts and subsequently converted to the logarithm of the minimal angle of resolution (logMAR) for analysis.
number of eyes with complications during and after surgery | within 18 months after surgery
  number of eyes with different complications such as shallow anterior chamber, malignant glaucoma,hyphema, Exudation in the anterior chamber,Corneal edema,Choroidal detachment,intraocular pressure spike on postoperative day 1

CONTACTS AND LOCATIONS:
Overall Officials: Jian Ge, MD, PhD, Principal Investigator — Zhongshan Ophthalmic Center, Sun Yat-sen University

REFERENCES:
- [Background] Gazzard G, Foster PJ, Devereux JG, Oen F, Chew P, Khaw PT, Seah S. Intraocular pressure and visual field loss in primary angle closure and primary open angle glaucomas. Br J Ophthalmol. 2003 Jun;87(6):720-5. doi: 10.1136/bjo.87.6.720. PMID 12770969
- [Background] Gelber EC, Anderson DR. Surgical decisions in chronic angle-closure glaucoma. Arch Ophthalmol. 1976 Sep;94(9):1481-4. doi: 10.1001/archopht.1976.03910040315004. PMID 962659
- [Background] Sihota R, Gupta V, Agarwal HC. Long-term evaluation of trabeculectomy in primary open angle glaucoma and chronic primary angle closure glaucoma in an Asian population. Clin Exp Ophthalmol. 2004 Feb;32(1):23-8. doi: 10.1046/j.1442-9071.2004.00752.x. PMID 14746586
- [Background] Hong S, Park K, Ha SJ, Yeom HY, Seong GJ, Hong YJ. Long-term intraocular pressure control of trabeculectomy and triple procedure in primary open angle glaucoma and chronic primary angle closure glaucoma. Ophthalmologica. 2007;221(6):395-401. doi: 10.1159/000107499. PMID 17947826
- [Background] Zhang X, Teng L, Li A, Du S, Zhu Y, Ge J. The clinical outcomes of three surgical managements on primary angle-closure glaucoma. Yan Ke Xue Bao. 2007 Jun;23(2):65-74. PMID 17867508
- [Background] Wang M, Ge J, Lin MK, Zhuo YH, Ling YL, Fang M, Liu X, Peng SX, Yu MB. [Clinical observation of trabeculectomy for primary angle closure glaucoma]. Zhonghua Yan Ke Za Zhi. 2009 Apr;45(4):338-43. Chinese. PMID 19575967
- [Background] Tsai HY, Liu CJ, Cheng CY. Combined trabeculectomy and cataract extraction versus trabeculectomy alone in primary angle-closure glaucoma. Br J Ophthalmol. 2009 Jul;93(7):943-8. doi: 10.1136/bjo.2008.151803. Epub 2009 Apr 20. PMID 19383599
- [Background] Wishart PK, Atkinson PL. Extracapsular cataract extraction and posterior chamber lens implantation in patients with primary chronic angle-closure glaucoma: effect on intraocular pressure control. Eye (Lond). 1989;3 ( Pt 6):706-12. doi: 10.1038/eye.1989.109. PMID 2630350
- [Background] Acton J, Salmon JF, Scholtz R. Extracapsular cataract extraction with posterior chamber lens implantation in primary angle-closure glaucoma. J Cataract Refract Surg. 1997 Jul-Aug;23(6):930-4. doi: 10.1016/s0886-3350(97)80255-6. PMID 9292680
- [Background] Gunning FP, Greve EL. Lens extraction for uncontrolled angle-closure glaucoma: long-term follow-up. J Cataract Refract Surg. 1998 Oct;24(10):1347-56. doi: 10.1016/s0886-3350(98)80227-7. PMID 9795850
- [Background] Hayashi K, Hayashi H, Nakao F, Hayashi F. Effect of cataract surgery on intraocular pressure control in glaucoma patients. J Cataract Refract Surg. 2001 Nov;27(11):1779-86. doi: 10.1016/s0886-3350(01)01036-7. PMID 11709251
- [Background] Liu CJ, Cheng CY, Wu CW, Lau LI, Chou JC, Hsu WM. Factors predicting intraocular pressure control after phacoemulsification in angle-closure glaucoma. Arch Ophthalmol. 2006 Oct;124(10):1390-4. doi: 10.1001/archopht.124.10.1390. PMID 17030705
- [Background] Tham CC, Kwong YY, Leung DY, Lam SW, Li FC, Chiu TY, Chan JC, Lam DS, Lai JS. Phacoemulsification versus combined phacotrabeculectomy in medically uncontrolled chronic angle closure glaucoma with cataracts. Ophthalmology. 2009 Apr;116(4):725-31, 731.e1-3. doi: 10.1016/j.ophtha.2008.12.054. Epub 2009 Feb 25. PMID 19243831
- [Background] Tham CC, Kwong YY, Leung DY, Lam SW, Li FC, Chiu TY, Chan JC, Chan CH, Poon AS, Yick DW, Chi CC, Lam DS, Lai JS. Phacoemulsification versus combined phacotrabeculectomy in medically controlled chronic angle closure glaucoma with cataract. Ophthalmology. 2008 Dec;115(12):2167-2173.e2. doi: 10.1016/j.ophtha.2008.06.016. Epub 2008 Sep 18. PMID 18801576
- [Background] Zhuo YH, Wang M, Li Y, Hao YT, Lin MK, Fang M, Ge J. Phacoemulsification treatment of subjects with acute primary angle closure and chronic primary angle-closure glaucoma. J Glaucoma. 2009 Dec;18(9):646-51. doi: 10.1097/IJG.0b013e31819c4322. PMID 20010241
- [Background] Wedrich A, Menapace R, Radax U, Papapanos P. Long-term results of combined trabeculectomy and small incision cataract surgery. J Cataract Refract Surg. 1995 Jan;21(1):49-54. doi: 10.1016/s0886-3350(13)80479-8. PMID 7722902
- [Background] Park HJ, Weitzman M, Caprioli J. Temporal corneal phacoemulsification combined with superior trabeculectomy. A retrospective case-control study. Arch Ophthalmol. 1997 Mar;115(3):318-23. doi: 10.1001/archopht.1997.01100150320002. PMID 9076202
- [Background] Kim JW, Jung CI, Hwang HS. Comparative study of three phacotrabeculectomy procedures through a single incision. Korean J Ophthalmol. 1998 Jun;12(1):30-6. doi: 10.3341/kjo.1998.12.1.30. PMID 9753949
- [Background] Wu WC, Wu SC, Lin SM. Surgical outcome of combined phacoemulsification and trabeculectomy. Changgeng Yi Xue Za Zhi. 1999 Dec;22(4):572-8. PMID 10695203
- [Background] Tow SL, Aung T, Oen FT, Seah SK. Combined phacoemulsification, intraocular lens implantation and trabeculectomy for chronic angle closure glaucoma. Int Ophthalmol. 2001;24(5):283-9. doi: 10.1023/a:1025478923950. PMID 14531631
- [Background] Kleinmann G, Katz H, Pollack A, Schechtman E, Rachmiel R, Zalish M. Comparison of trabeculectomy with mitomycin C with or without phacoemulsification and lens implantation. Ophthalmic Surg Lasers. 2002 Mar-Apr;33(2):102-8. PMID 11942540
- [Background] Lai JS, Tham CC, Chan JC, Lam DS. Phacotrabeculectomy in treatment of primary angle-closure glaucoma and primary open-angle glaucoma. Jpn J Ophthalmol. 2004 Jul-Aug;48(4):408-11. doi: 10.1007/s10384-003-0075-2. PMID 15295672
- [Background] Zarei R, Azimi R, Moghimi S, Abdollahi A, Amini H, Eslami Y, Fakhraii G. Inhibition of intraocular fibrin formation after infusion of low-molecular-weight heparin during combined phacoemulsification-trabeculectomy surgery. J Cataract Refract Surg. 2006 Nov;32(11):1921-5. doi: 10.1016/j.jcrs.2006.06.029. PMID 17081897
- [Background] Cantor LB, Mantravadi A, WuDunn D, Swamynathan K, Cortes A. Morphologic classification of filtering blebs after glaucoma filtration surgery: the Indiana Bleb Appearance Grading Scale. J Glaucoma. 2003 Jun;12(3):266-71. doi: 10.1097/00061198-200306000-00015. PMID 12782847